CLINICAL TRIAL: NCT07231874
Title: Preservation of the Alveolar Ridge Using a Cortical Lamina After Tooth Extraction: A Randomized Controlled Clinical Trial
Brief Title: Cortical Lamina for Alveolar Ridge Preservation
Acronym: Lamina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/01
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-01

CONDITIONS: Tooth Extraction; Periapical Infections; Tooth Fracture; Periodontal Disease, AVDC Stage 4; Hopeless Tooth
Keywords: ridge preservation; Cortical Lamina; Bone Regeneration; Alveolar Bone Loss; Tooth extraction; Implant Site Development; Buccal Bone
MeSH Terms: conditions — Tooth Fractures; Periodontal Diseases; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. In the test group, a cortical lamina will be placed between the elevated mucoperiosteal flap and the buccal bone plate immediately after tooth extraction. In the control group, extraction sockets will heal spontaneously without lamina placement. Both groups will be followed for six months before implant placement to assess dimensional changes in the alveolar ridge.
Who Masked: Outcomes Assessor
Masking Description: Participants and surgeons will know group allocation; however, the radiographic examiner assessing outcomes will remain blinded to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group - Cortical Lamina Placement (Experimental): Following atraumatic tooth extraction, a small full-thickness flap will be elevated without releasing incisions. A cortical lamina will be placed between the buccal bone plate and the elevated flap to isolate the periosteum and stabilize the ridge contour. The flap will then be repositioned and sutured for non-submerged healing. Sutures will be removed after two weeks. Standard postoperative care will include 0.12% chlorhexidine mouth rinses and analgesics as needed.
  Interventions: Procedure: Cortical Lamina Technique
- Control Group - Spontaneous Healing (Active Comparator): After tooth extraction, the site will be allowed to heal naturally without the placement of cortical lamina or any grafting material. The flap will be repositioned and sutured for non-submerged healing. Postoperative care will follow the same protocol as the test group.
  Interventions: Procedure: Natural Healing (Control)

INTERVENTIONS:
Procedure: Cortical Lamina Technique — Surgical placement of a cortical lamina between the buccal bone plate and elevated mucoperiosteal flap immediately after tooth extraction. The lamina serves as a barrier to stabilize the alveolar contour and promote bone preservation. The flap is sutured for non-submerged healing, and postoperative care includes chlorhexidine rinses and analgesics as needed.
  Arms: Test Group - Cortical Lamina Placement
Procedure: Natural Healing (Control) — After tooth extraction, the site will heal naturally without placement of cortical lamina or any grafting material. The flap is repositioned and sutured for non-submerged healing. Postoperative care is identical to the test group.
  Arms: Control Group - Spontaneous Healing

SUMMARY:
This randomized controlled clinical trial aims to evaluate the efficacy of placing a cortical lamina between the elevated flap and buccal bone plate following tooth extraction for preserving alveolar ridge dimensions. Forty patients will be randomly assigned to either the test group (lamina placement) or control (no intervention). Changes in ridge width and height will be assessed using CBCT and 3D digital models after six months.

DETAILED DESCRIPTION:
Alveolar bone resorption after tooth extraction can compromise prosthetic and implant rehabilitation by reducing both bone height and width, especially at the buccal plate. Various alveolar ridge preservation (ARP) techniques have been proposed to minimize these dimensional changes; however, their clinical predictability and long-term benefit remain debated.

This randomized controlled clinical trial aims to evaluate the efficacy of placing a cortical lamina between the elevated mucoperiosteal flap and the buccal bone plate immediately after tooth extraction to preserve alveolar ridge dimensions. The technique is intended to limit post-extraction resorption by temporarily isolating the periosteum from the underlying bone, promoting favorable bone remodeling and contour maintenance for subsequent implant placement.

Forty patients requiring the extraction of single teeth (premolars, canines, or maxillary incisors) will be enrolled and randomly allocated into two groups:

Test group: A cortical lamina will be inserted between the buccal bone and the flap following tooth extraction.

Control group: Extraction sites will be left untreated to heal spontaneously.

All surgeries will be performed under local anesthesia by calibrated clinicians. Healing will occur by primary intention without submerged flaps. Sutures will be removed after two weeks. Patients will follow standardized postoperative care, including chlorhexidine rinses and analgesics as needed.

Cone-beam computed tomography (CBCT) and digital impressions will be obtained at baseline (immediately post-extraction) and at six months. The primary outcome is the linear change in ridge width and height measured on CBCT scans. Secondary outcomes include volumetric dimensional changes analyzed from 3D digital impressions.

Data will be analyzed using parametric or non-parametric tests depending on normal distribution (ANOVA or Kruskal-Wallis, with appropriate post-hoc comparisons). A significance level of p < 0.05 will be applied.

The study follows the Declaration of Helsinki and CONSORT 2010 guidelines. Ethical approval has been granted by the Comité de Ética de la Investigación, Universidad de Ciencias Médicas de La Habana (Aval 2024/01, April 9 2024).

ELIGIBILITY:
Inclusion Criteria:

* Presence of a tooth indicated for extraction (maxillary incisors, canines, or premolars in either jaw).
* Age ≥ 21 years.
* Good general health with no contraindications for oral surgery.
* Non-pregnant individuals.
* Willingness to participate and sign written informed consent.

Exclusion Criteria:

* Uncontrolled systemic disease (e.g., diabetes mellitus, hypertension).
* History of chemotherapy or radiotherapy.
* Current smokers of more than 10 cigarettes per day.
* Sites previously treated with regenerative or augmentation procedures.
* Poor oral hygiene or active periodontal infection.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Alveolar Ridge Width and Height | Baseline (immediately post-extraction) to 6 months after extraction
  Linear dimensional changes in the alveolar ridge (horizontal width and vertical height) will be evaluated using cone-beam computed tomography (CBCT) images taken immediately after tooth extraction (baseline) and six months post-surgery. Measurements will be made at standardized reference points on cross-sectional CBCT slices to quantify resorption or preservation of bone.

SECONDARY OUTCOMES:
Volumetric Change of the Alveolar Ridge | Baseline to 6 months post-extraction
  Volumetric dimensional changes of the alveolar ridge will be assessed by comparing 3D digital models of the extraction sites obtained from intraoral impressions taken at baseline (immediately post-extraction) and six months after surgery. Superimposition and digital analysis will be performed to quantify total volume loss or preservation of the alveolar ridge contour.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Sciences of Havana, Havana, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted at a single clinical center with a limited sample size, and the data contain identifiable clinical imaging and patient information. Aggregated results and summary analyses will be made available through scientific publications and conference presentations.

REFERENCES:
- [Result] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Result] Atieh MA, Alsabeeha NH, Payne AG, Duncan W, Faggion CM, Esposito M. Interventions for replacing missing teeth: alveolar ridge preservation techniques for dental implant site development. Cochrane Database Syst Rev. 2015 May 28;2015(5):CD010176. doi: 10.1002/14651858.CD010176.pub2. PMID 26020735
- [Result] Richardson CR, Mellonig JT, Brunsvold MA, McDonnell HT, Cochran DL. Clinical evaluation of Bio-Oss: a bovine-derived xenograft for the treatment of periodontal osseous defects in humans. J Clin Periodontol. 1999 Jul;26(7):421-8. doi: 10.1034/j.1600-051x.1999.260702.x. PMID 10412845
- [Result] Lee JH, Yi GS, Lee JW, Kim DJ. Physicochemical characterization of porcine bone-derived grafting material and comparison with bovine xenografts for dental applications. J Periodontal Implant Sci. 2017 Dec;47(6):388-401. doi: 10.5051/jpis.2017.47.6.388. Epub 2017 Dec 31. PMID 29333325
- [Result] Klinge B, Alberius P, Isaksson S, Jonsson J. Osseous response to implanted natural bone mineral and synthetic hydroxylapatite ceramic in the repair of experimental skull bone defects. J Oral Maxillofac Surg. 1992 Mar;50(3):241-9. doi: 10.1016/0278-2391(92)90320-y. PMID 1311759
- [Result] Al Qabbani A, Al Kawas S, A Razak NH, Al Bayatti SW, Enezei HH, Samsudin AR, Sheikh Ab Hamid S. Three-Dimensional Radiological Assessment of Alveolar Bone Volume Preservation Using Bovine Bone Xenograft. J Craniofac Surg. 2018 Mar;29(2):e203-e209. doi: 10.1097/SCS.0000000000004263. PMID 29303859